CLINICAL TRIAL: NCT02138643
Title: Laparoscopy Heller Myotomy With Fundoplication Associated Versus Peroral Endoscopic Myotomy (POEM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23460613000000068
Record Dates: First submitted 2014-04-16; First posted 2014-05-14 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Dysphagia; Achalasia
Keywords: Achalasia; Megaesophagus; Peropal endoscopic myotomy(POEM); Laparoscopic Heller myotomy
MeSH Terms: conditions — Deglutition Disorders; Esophageal Achalasia | interventions — Endoscopy; Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endoscopic surgery (Active Comparator): Patients with symptomatic achalasia confirmed by clinical and laboratory tests, which meet the criteria for inclusion and exclusion. These will be treated with Endoscopic surgery - Peroral endoscopic myotomy (POEM)
  Interventions: Procedure: Endoscopic surgery
- Laparoscopic surgery (Sham Comparator): Patients with symptomatic achalasia confirmed by clinical and laboratory tests, which meet the criteria for inclusion and exclusion. These will be treated with Laparoscopic surgery - Laparoscopic Heller myotomy.
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Endoscopic surgery — These will be treated with Endoscopic surgery - Peroral endoscopic myotomy (POEM)
  Arms: Endoscopic surgery
Procedure: Laparoscopic surgery — These will be treated with Laparoscopic surgery - Laparoscopic Heller myotomy.
  Arms: Laparoscopic surgery

SUMMARY:
Achalasia is a disorder benign esophageal motor, which is characterized by failure to relax the lower esophageal sphincter ( LES) in response to swallowing associated with lack of peristalsis of the esophageal body. Its most common clinical presentation is dysphagia , and occasionally chest pain , regurgitation , aspiration pneumonia and weight loss , resulting in a large impact on daily activities and quality of life of affected individuals .

There is currently considered curative treatment for achalasia , dysphagia relief being the primary therapeutic target and is forced to relax the LES by endoscopy or surgery. Thus , the most commonly used endoscopic treatments are forced dilatation of the cardia and botulinum toxin. Laparoscopic Heller myotomy with antireflux procedure with therapy is considered "gold standard " because of excellent results and minimal invasiveness. Currently , pneumatic dilation and surgical treatment with the Heller myotomy with fundoplication are strongly associated with the best therapeutic options available .

In recent years, the possibility of using endoluminal access in the treatment of achalasia patients through the technique originally described as Natural orifices Translumenal Endoscopic Surgery ( NOTES) and continuing advances in the submucosal dissection has enabled the concomitant development of a new approach described as perioral endoscopic myotomy . In 2007, Pasricha et al , described the feasibility of endoscopic esophageal myotomy through a submucosal tunnel initially in an animal model . The first performance of this procedure in humans was described by Inoue et al , in 2010 , introducing the concept of transluminal endoscopic surgery through natural orifices , with the objective of minimizing the trauma and all the stress resulting from open surgical procedure . These authors call the procedure as POEM ( Per Oral Endoscopic myotomy ) .

DETAILED DESCRIPTION:
Achalasia is a disorder benign esophageal motor, which is characterized by failure to relax the lower esophageal sphincter ( LES) in response to swallowing associated with lack of peristalsis of the esophageal body . Its most common clinical presentation is dysphagia , and occasionally chest pain , regurgitation , aspiration pneumonia and weight loss , resulting in a large impact on daily activities and quality of life of affected individuals .

Epidemiological data show an incidence in the United States and Europe , approximately 1/200.000 and no predilection for sex, age group (mean between 25 and 60 years) was observed , as well as any other demographic group . In Brazil , the incidence is approximate 7-13/100.000 inhabitants .

Large proportion of patients with symptomatic achalasia require additional tests for diagnosis. Endoscopy ( EDA ) despite being regarded as a major test for initial evaluation of dysphagia , presents serious limitations to evaluate esophageal motility , especially in early stages . Some contrast studies , highlighting the Esophagogram barium ( DSE ) , provide additional anatomical findings as esophageal shape and size , as well as functional : peristalsis , the LES function and bolus clearance through the esophagogastric junction ( TEG ) . Another useful method of diagnosis is the Esophageal manometry , with characteristic (Chicago Classification of Distal Esophageal Motility Disorders ) : aperistalsis the esophageal body and failure to relax the LES , currently best characterized by High Resolution Manometry .

Idiopathic achalasia is confined to the esophagus and has no established etiology , with agenesis of the myenteric plexus or viral infections , in particular herpes simplex ( HSV - 1 ) , the most likely hypothesis . In Brazil , the secondary achalasia caused by Chagas disease predominantly among other etiologies , involves but is expressed primarily systemic disease with esophageal involvement . Infected patients Typanossoma cruzi, the causative agent of Chagas disease , 7-10 % have esophageal involvement, and due to its chronic nature the most common clinical presentation is megaesophagus , to varying degrees .

There is currently considered curative treatment for achalasia , dysphagia relief being the primary therapeutic target and is forced to relax the LES by endoscopy or surgery . Thus , the most commonly used endoscopic treatments are forced dilatation of the cardia and botulinum toxin. Laparoscopic Heller myotomy with antireflux procedure with therapy is considered "gold standard " because of excellent results and minimal invasiveness . Currently , pneumatic dilation and surgical treatment with the Heller myotomy with fundoplication are strongly associated with the best therapeutic options available .

Many studies have validated the efficacy of pneumatic dilation in some cases exceeding 90%, but with the limitation of the need for serial dilations , the main complication being perforation , around 8 % .

With the introduction of minimally invasive surgery , surgical approach has gained great clinical importance , especially for laparoscopic Heller myotomy with antireflux valve ( fundoplication ) . With a success rate ranging between 89 and 100 % in recent studies , provide a more lasting relief of symptoms without the need for additional interventions , compared to pneumatic dilation .

In recent years, the possibility of using endoluminal access in the treatment of achalasia patients through the technique originally described as Natural orifices Translumenal Endoscopic Surgery ( NOTES) and continuing advances in the submucosal dissection has enabled the concomitant development of a new approach described as perioral endoscopic myotomy . In 2007, Pasricha et al , described the feasibility of endoscopic esophageal myotomy through a submucosal tunnel initially in an animal model . The first performance of this procedure in humans was described by Inoue et al , in 2010 , introducing the concept of transluminal endoscopic surgery through natural orifices , with the objective of minimizing the trauma and all the stress resulting from open surgical procedure . These authors call the procedure as POEM ( Per Oral Endoscopic myotomy ) .

OBJECTIVE The primary objective of this protocol is to compare the efficacy between surgical approach through laparoscopic myotomy with fundoplication associated Heller myotomy and endoscopic peroral ( POEM ) in the treatment of patients with achalasia regardless of its etiology .

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years diagnosed with symptomatic achalasia (dysphagia score ≥ II and Eckardt> 3) all grades including Rezende classification and Chicago Classification.
* Patients who agree to participate in the study and signed an informed consent.

Exclusion Criteria:

* Treatment (s) prior (s) achalasia.
* Patients with a history of esophageal, mediastinal and / or gastric surgery (except for gastric perforation).
* Patients with liver cirrhosis and / or esophageal varices, Barrett's esophagus, esophageal stricture, premalignant or malignant esophageal lesions and coagulopathy.
* Patients with severe cardiopulmonary disease or other serious illness that results in a high surgical risk.
* Patients diagnosed with pseudoachalasia
* Patients diagnosed with diverticulum in the distal esophagus.
* Pregnancy and lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Remission of symptoms dysphagia. | 12 months after the procedure performed.
  Patient selection will last for six months after the beginning of the study. Six months later, conduct additional examinations and randomization. Twelve months after the start of the project will be the completion of endoscopic surgery or laparoscopic surgery for resolution of dysphagia. The measure is a composite.

SECONDARY OUTCOMES:
Running time of the procedure and hospitalization. | Starts 12 months after procedure performed.
  New outpatient medical visits for clinical reassessment, more precisely 30 days, 3 months, 6 months and 12 months after the procedure will be scheduled to measure the execution time of the procedure and hospitalization. The measure is a composite.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Sakai, Principal Investigator — Hospital das Clínicas da FMUSP; Eduardo Turiani H de Moura, Study Director — Hospital das Clínicas FMUSP
Locations (1):
- Hospital das Clínicas da FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No